CLINICAL TRIAL: NCT04874740
Title: Seroprevalence of the Anti-SARS-CoV-2 Antibodies in Kidney Transplant Recipients in Severely Affected Region
Brief Title: Seroprevalence of the Anti-SARS-CoV-2 Antibodies (Causing COVID-19) in Kidney Transplant Recipients in Severely Affected Region
Acronym: SECOVtx
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: 2/IK-FNO/2021
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: COVID-19 Pandemic; Transplantation, Kidney
Keywords: COVID-19; Seroepidemiologic Studies; Kidney transplant
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipients: Collection of data from kidney transplant patients at regular outpatient check-ups.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Goal of this study is to evaluate the seroprevalence of anti-SARS-CoV-2 antibodies in patients after kidney transplantation who are one of the risk groups for the severe course of the infection and map the progression of the virus throughout this specific part of population, which is also important for possible future epidemics. We will evaluate the seroprevalence of anti-SARS-CoV-2 antibodies according to age and gender. We will compare seroprevalence in all measured antibodies types and we will also assess the development of antibodies level in positive patients.

DETAILED DESCRIPTION:
The Czech Republic (Central Europe region) is one of the most affected countries in the World by COVID 19 pandemic. By 1st of March 2021, the SARS-COV-2 virus infection was proven in the Czech Republic in 1 247 051 thousand people, which is 11.7% of the population (11 627 per 100 000, in the USA 8743/100 000, in the UK 6300/100 000, in the Germany 2879/100 000, France 5379/100 000). The rapidly increasing number of people infected in October 2020 have led to adoption of strict countrywide epidemic measures, which are still largely ongoing. During first 2 months of 2021 was still serious spread of the virus in population with increasing numbers of infected persons.

The SARS-CoV-2 virus can be detected in the body by several ways. The presence of the virus can be directly confirmed by RT-PCR or by determination of viral antigen from a swab from the nasopharynx, throat, direct examination of sputum or aspirate from bronchoscopy, or rectum. Indirect methods of virus detection include the determination of antibodies in the blood. Antibodies can target several structures of the virus: spike protein (S), envelope, membrane or nucleocapsid (NP). The S protein is composed of S1 and S2 subunit. The S1 subunit contains receptor-binding domain (RBD) which is necessary for interaction and entering human cells. In practice, IgG, IgM and IgA antibodies against RBD and NP are usually detected.2,3 With regard of serious development of the COVID 19 epidemic situation in the Czech Republic, we decided to do this prevalence study. Our goal is to evaluate the seroprevalence of anti-SARS-CoV-2 antibodies in patients after kidney transplantation which is also important for possible future epidemics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Recipient of a transplanted kidney
* Planned visit to the outpatient nephrology clinic of University Hospital Ostrava, Czech Republic, between 1.5. and 30.7.2021 for enrolment
* Planned blood collection and available results of blood tests from planned inspections from 18.1.2021.
* Signed consent to the use of anonymous data for scientific purposes and publications.

Exclusion Criteria:

* disagreement with participation in the study and data analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after any kidney transplantation, monitored regularly in the nephrology clinic of the University Hospital Ostrava.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with positive anti-SARS-CoV-2 antibodies (one or more) | Between 18 January 2020 and 30 September 2022
  Seroprevalence of anti-SARS-Cov 2 antibodies - in how many patients is positive at least one of the measured antibodies against SARS-Cov-2 virus (IgA, IgM or IgG against RBD, IgG against nucleocapsid).

SECONDARY OUTCOMES:
Number od Participants with change of baseline of anti-SARS-COV-2 antibodies | From May 1, 2021 to September 30, 2022
  Development of antibodies in the observed period during follow up.
Number of Participants with positive anti-SARS-COV-2 antibodies in groups divided by age, sex, blood type. | Between 18 January 2020 and 30 September 2022
  Seroprevalence depending on age, sex, blood type, time of measurement, time since transplantation, residence, type of immunosuppression.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vaclavik, prof.,M.D., Study Chair — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: Undecided